CLINICAL TRIAL: NCT04565548
Title: Effect of an Educational Program for Hypertensive Patients: a Randomized Controlled Trial
Brief Title: Hypertension Treatment Adherence Improving Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HSEARS20200821002
Record Dates: First submitted 2020-09-10; First posted 2020-09-25 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2020-09

CONDITIONS: Hypertension,Essential
Keywords: hypertension; adherence; self-efficacy; educational intervention
MeSH Terms: conditions — Essential Hypertension; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will not participate in group allocation or intervention delivery.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will receive the newly developed theory-guided program for 12 weeks.
  Interventions: Other: Educational program for hypertensive patients
- Control (Active Comparator): Participants will receive the usual care and non-hypertension related text messaging for 12 weeks.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Educational program for hypertensive patients — The theory-guided program consisted of one session of health education, self-developed leaflet, and weekly text messaging for 12 weeks.
  Arms: Intervention
Other: Usual care — One standardized health education and a leaflet developed by the Health Bureau. As similar as the intervention group, weekly text messaging will be delivered, but the content is not related to the blood pressure control.
  Arms: Control

SUMMARY:
Persistent adherence to lifestyle modifications and blood pressure lowering medications were the best way to control blood pressure. But low adherence was noted in reviews and studies resulting those taking blood pressure lowering medications could not achieve a controlled blood pressure. In this study, a theory-guided educational program will be developed with an aim to improve the blood pressure, self-efficacy and adherence behaviors among those diagnosed with high blood pressure in the community. 148 participants will be recruited and divided into control group and intervention group randomly in a ratio of 1:1. The intervention group will receive the theory-guided educational program, while the control group will receive the usual care. The study will last for 12 weeks. Data will be collected at baseline, week 8 and week 12. SPSS and generalized estimating equations model will be employed for data analysis. The results will inform an effective way to conduct health promotion in community. The improved adherence to lifestyle modifications and medications will be beneficial to the clients' health.

DETAILED DESCRIPTION:
Persistent adherence to lifestyle modifications and anti-hypertensive medications were emphasized in hypertension guidelines to control blood pressure effectively. But low adherence to lifestyle modifications and medication were noted in reviews and studies. Low adherence would lead to those received hypertension treatment did not achieve a controlled blood pressure. In this study, an educational program guided by the Health Promotion Model will be conducted to examine the effect on blood pressure, self-efficacy and treatment adherence among hypertensive patients in the community. A 2-arm parallel randomized control trial will be conducted. 148 participants will be recruited and divided into control and intervention group in a ration of 1:1. The intervention group will receive the theory-guided educational program, while the control group will receive the usual care. The study will last for 12 weeks. Data will be collected at baseline, week 8 and week 12. SPSS and generalized estimating equations model will be employed for data analysis. The results will inform community healthcare professionals about the effective way for health promotion, to enhance the adherence to lifestyle modifications and medications among hypertensive clients resulting sustainable benefits to the clients' health.

ELIGIBILITY:
Inclusion Criteria:

* Own a mobile phone and able to use
* Able to communicate with Cantonese and read Chinese
* Diagnosed with hypertension and taking at least one anti-hypertensive medication
* SBP = 131~159 mmHg or DBP = 81~99 mmHg

Exclusion Criteria:

* Renal hypertension
* Mini-Cog < 3

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2021-03-06 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change of blood pressure at week 8 and week 12 | Baseline, week 8, week 12
  Systolic and diastolic blood pressure (mmHg) is measured by a trained research assistant. A validated upper-arm blood pressure monitor is used for the blood pressure measurement.

SECONDARY OUTCOMES:
Change of Treatment Adherence Questionnaire for Patients with Hypertension (TAQPH) at week 8 and week 12 | Baseline, week 8, week 12
  TAQPH consists of 28 items and covers the adherence to medications and lifestyle modifications in hypertension management. The responses are made on a 1-4 scale, and the sum of the score ranges from 28 to 112. The TAQPH has been proved to be reliable with good Cronbach's alpha coefficient 0.86 for Chinese hypertensive adults.
Change of Self-efficacy for managing chronic disease (SEMCD) at week 8 and week 12 | Baseline, week 8, week 12
  SEMCD consists of six self-report items to measure the self-efficacy of hypertension management. Summative scores range from 6 to 60. The scale was translated into Chinese and yielded a good reliability (Cronbach's alpha = 0.88-0.98; teste-retest reliability = 0.73-0.98) in Chinese hypertensive adults and Chinese older adults.

CONTACTS AND LOCATIONS:
Overall Officials: Eliza Mi Ling Wong, Dr, Principal Investigator — The Hong Kong Polytechnic University
Locations (2):
- Community Health Centres, Shenzhen, Shenzhen, China
- Complexo de Apoio à Família e de Serviço Comunitário de Seac Pai Van da União Geral das Associações dos Moradores de Macau, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tam HL, Wong EML, Cheung K. Educational Program with Text Messaging for Community-Dwelling Patients with Hypertension: A Pilot Randomized Controlled Trial. Asian Nurs Res (Korean Soc Nurs Sci). 2023 Aug;17(3):158-166. doi: 10.1016/j.anr.2023.06.001. Epub 2023 Jun 7. PMID 37295501